CLINICAL TRIAL: NCT03666130
Title: Endoscopic Versus Conventional Septoplasty in the Treatment of Deviated Nasal Septum
Brief Title: Endoscopic Versus Conventional Septoplasty in Treatment of Deviated Nasal Septum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahrous, Institutional Review Board (IRB) of faculty of medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: septoplasty of DNS
Record Dates: First submitted 2018-07-30; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Endoscopic Septoplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic septoplasty (Active Comparator): in this arm the participants will undergo endoscopic septoplasty for correction of the deviated nasal septum
  Interventions: Procedure: endoscopic septoplasty
- conventional septoplasty (Active Comparator): in this arm the participants will undergo conventional septoplasty operation for correction of the deviated nasal septum that will done by surgical traditional septoplasty technique using head lamb and anterior rhinoscopy
  Interventions: Procedure: endoscopic septoplasty

INTERVENTIONS:
Procedure: endoscopic septoplasty — endoscopic septoplasty is the use of nasal endoscopy in the septoplasty surgery for treatment of deviated nasal septum . we aim to compare the outcome of using this method versus conventional septoplasty

SUMMARY:
This study aims to compare the two techniques of relieving nasal obstruction, and its efficacy in the relief of headache, hyposmia and post-nasal drip and nasal synechiae formation and /or other postoperative complications following each techniques of surgery.

DETAILED DESCRIPTION:
A straight septum is found not to be the dominant but the exception.

A deviated septum can be asymptomatic or can cause functional and cosmetic abnormality. it also can become symptomatic at any age. Deviated nasal septum not only causes breathing difficulties but also causes improper aeration of para nasal sinuses leading to infection, so any functional or cosmetic disturbance caused by a deviated septum should be treated. Different surgeries have been proposed for the correction of deviated nasal septum. Initially, submucosal resection of septum was proposed but was later replaced by septoplasty .

Septoplasty is the procedure of choice in nasal obstruction caused by septal deviation resistant to medical treatment. It also improves access to the medial meatus in sinus surgery and other nasal and sinus procedures, such as cosmetic rhinoplasty and functional endoscopic sinus surgery(FESS)

Modern septoplasty techniques were initially described separately in the early twenties century by Killian and Freer. It is conventionally performed under direct visualization using a headlight and nasal speculum. However, this method has the drawbacks of relatively poor illumination and accessibility and no magnification, calling for a larger incision and elevation of larger flaps often on both sides of the septum. As a result, there are higher chances of over-resection and over manipulation. Endoscopic septoplasty has been commonly performed since the development of endonasal surgery and as as an alternative to the conventional technique. In this study the I investigators aim to compare the two techniques of relieving nasal obstruction, and its efficacy in the relief of headache, hyposmia and post-nasal drip and nasal synechiae formation following each techniques of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with deviated nasal septum with persistent symptoms for at least 3 months and had not responded to maximal medical management.
* patients of deviated nasal septum cased by either childbirth trauma or recent

Exclusion Criteria:

1. patients of asymptomatic deviated nasal septum
2. patients who had a history of previous nasal surgery
3. patients who had other causes of nasal obstruction
4. patients who had received radiotherapy of head and neck region.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients free from symptoms after surgery | 3 months
  the relive of the nasal obstruction symptoms as difficult breathing and nasal discharge and the complication of each method of surgery as synechia formation and postoperative bleeding

REFERENCES:
- [Result] Clark DW, Del Signore AG, Raithatha R, Senior BA. Nasal airway obstruction: Prevalence and anatomic contributors. Ear Nose Throat J. 2018 Jun;97(6):173-176. doi: 10.1177/014556131809700615. PMID 30036414
- [Result] Chandra RK. Endoscopic septoplasty: "How I do it". Am J Rhinol Allergy. 2017 Jul 1;31(4):276-277. doi: 10.2500/ajra.2017.31.4436. PMID 28716180
- [Result] Hong CJ, Monteiro E, Badhiwala J, Lee J, de Almeida JR, Vescan A, Witterick IJ. Open versus endoscopic septoplasty techniques: A systematic review and meta-analysis. Am J Rhinol Allergy. 2016 Nov 1;30(6):436-442. doi: 10.2500/ajra.2016.30.4366. PMID 28124656
- [Result] Shah J, Roxbury CR, Sindwani R. Techniques in Septoplasty: Traditional Versus Endoscopic Approaches. Otolaryngol Clin North Am. 2018 Oct;51(5):909-917. doi: 10.1016/j.otc.2018.05.007. Epub 2018 Jul 17. PMID 30025848
- [Result] Sathyaki DC, Geetha C, Munishwara GB, Mohan M, Manjuanth K. A comparative study of endoscopic septoplasty versus conventional septoplasty. Indian J Otolaryngol Head Neck Surg. 2014 Jun;66(2):155-61. doi: 10.1007/s12070-013-0692-0. Epub 2013 Nov 24. PMID 24822154
- [Result] Skitarelic NB, Vukovic K, Skitarelic NP. Comparative evaluation of conventional versus endoscopic septoplasty for limited septal deviation and spur. J Laryngol Otol. 2009 Aug;123(8):939-40; author reply 940. doi: 10.1017/S0022215109005556. Epub 2009 May 27. No abstract available. PMID 19470189
- [Result] Atan D, Ozcan KM, Gurbuz AB, Dere H. The Effect of Septoplasty on Voice Performance in Patients With Severe and Mild Nasal Septal Deviation. J Craniofac Surg. 2016 Jul;27(5):1162-4. doi: 10.1097/SCS.0000000000002794. PMID 27380579
- [Result] Champagne C, Ballivet de Regloix S, Genestier L, Crambert A, Maurin O, Pons Y. Endoscopic vs. conventional septoplasty: A review of the literature. Eur Ann Otorhinolaryngol Head Neck Dis. 2016 Feb;133(1):43-6. doi: 10.1016/j.anorl.2015.11.004. Epub 2015 Dec 8. PMID 26679230